CLINICAL TRIAL: NCT02751125
Title: Jaw Bone Reconstruction Using a Combination of Autologous Mesenchymal Stem Cells and Biomaterial Prior to Dental Implant Placement
Brief Title: Reconstruction of Jaw Bone Using Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: University of Ulm (Other); Haukeland University Hospital (Other); Université de Nantes (Other)
Responsible Party: Principal Investigator, Cecilie Gjerde, Assosiate Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003139-50
Record Dates: First submitted 2016-03-22; First posted 2016-04-26 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Bone Atrophy
Keywords: Mesenchymal stem cells; bone augmentation; bone regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Augmentation of new alveolar bone (Experimental): Augmentation of atrophied alveolar ridge with mesenchymal stem cells( MSC) and bis calcium phosphate(BCP)
  Interventions: Drug: BCP with autologous mesenchymal stem cells (MSC).

INTERVENTIONS:
Drug: BCP with autologous mesenchymal stem cells (MSC). — Augmentation of narrow alveolar ridge with BCP and MSC
  Other Names: MSC and BCP

SUMMARY:
This pilot study is aimed to reconstruct atrophied posterior alveolar mandibular ridges using biomaterial and autologous bone marrow derived stem cells (BMMSC) and to insert an implant into the new bone in a prosthetically guided position.

DETAILED DESCRIPTION:
Eleven patients presenting with the need of an implant retained restoration in the posterior mandibula and an alveolar ridge of maximum 4.5 mm width.

A clinical examination, x- rays and Cone Beam CT(CBCT) are accessed. A sample of the patients' bone marrow is extracted from the posterior alveolar ridge, immediately shipped to the collaborating good clinical practice (GCP) cell laboratory for cell expansion, and returned after 21 days. The stem cells mixed with Bi Calcium Phosphate (BCP) are then used to augment the alveolar ridge. The material is covered with a titanium reinforced membrane before closure of the site. After four to six months a bone biopsy is performed and implants are installed in the regenerated bone.

The patient will be followed after 1, 2, 3, and 5 years where implant stability will be assessed. Furthermore the new formed bone will be clinically and radiologically assessed at the same time.

ELIGIBILITY:
Inclusion Criteria:Patients presenting with an indication for an implant and wanting implant-borne prosthetic restoration.

* Patients presenting with lateral or vertical bone loss (focusing lateral bone loss) of the mandible behind the canine tooth.
* Lateral (width 5 mm or less) bone loss preventing the insertion of an implant without prior bone augmentation.
* Endentate for more than 6 months in the region requiring reconstruction.
* Endentate concerning at least 2 missing teeth in the region requiring reconstruction.
* Absence of clinical signs of infection in the region requiring reconstruction.
* Patients presenting with good dental hygiene (subjective criteria)
* Patients not presenting with any major oral pathologies.
* Dental crest size less than 5 mm.

General criteria:

* Adult patients over 18 and under 80 years of age.
* Patients in good general health presenting with a complete blood count and renal and hepatic function values within normal limits (confirmed by local laboratory tests).
* Patients with the capacity to understand medical information and give their informed consent.

Exclusion Criteria:

ocal criteria:

* Patients presenting with clinical or radiological signs of bone infection (acute or chronic osteomyelitis).
* Residual dentition close to the area requiring reconstruction with untreated endodontic disorder (apical granuloma or apical cyst).
* Untreated oral infection (cellulitis, periodontitis).
* Patients with poor hygiene (subjective criteria).
* Surgical procedure undertaken in the area requiring reconstruction less than 6 months prior to the bone graft.
* History of malignant tumors of the upper airways / digestive tract or of the jaw.
* History of or scheduled cervico-facial radiation therapy.

General criteria:

* The patient suffers from any serious coagulation disorders that could require substitution therapy
* The patient is receiving VKA therapy, which should be adjusted if necessary so that the INR does not exceed 2.5
* The patient has history of allergy to iodine or to local anesthetics(sulfites, etc.)., or a history of hematoma, or hemorrhage or blood coagulation disorders
* The patient has received localized iliac crest radiotherapy contraindicating withdrawal from the irradiated site
* The patient has major skin lesions or diseases.
* Patients presenting with bone metabolism disorders: hypophosphatemia, primary parathyroid osteitis or that is secondary to chronic renal insufficiency or osteomalacia, Paget's disease, vitamin D-related disorders, osteoporosis.
* Pregnant or breastfeeding women or women not using effective contraception if they are of childbearing age.
* Patients presenting with cancerous disorders (carcinoma, sarcoma, leukemia, lymphoma) or psychiatric disorders or with uncontrolled systemic diseases (diabetes, hypertension), or chronic renal disease.
* Severe bruxism.
* History of chemotherapy.
* Smoking or alcohol addiction. Occasional consumption of alcohol and/or smoking will be noted in the case report form.
* Patients with an ASA score of 0 or 1, incapable of tolerating general anesthesia.
* Immunosuppression
* Body mass index outside the normal range, particularly >30 because of increased surgical risk at the time of BM harvesting from the iliac crest.
* Risk of remote infection (orthopedic prosthesis implanted in the previous 6 months, patients presenting with a high risk of infective endocarditis, presence of pulmonary arteriovenous shunt, etc.).
* HIV, HTLV and/or syphilis seropositivity.
* Hepatitis B or C infection.
* Active autoimmune disease.
* History of immunosuppressant treatment or bone marrow treatment.
* Administration of treatment interfering with bone metabolism.
* Patients requiring antibiotic prophylaxis before any dental procedure
* Patients reticent to undergo dental care or periodontal treatment
* Concomitant treatments: history of treatment or current treatment with bisphosphonates, long term corticosteroid treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Amount of newly formed bone induced by MSCs and the bone substitute. These measurements are based on radiological assessments. | Four to six months post augmentation
  CBCT

SECONDARY OUTCOMES:
Implant stability | 12 months
  Implant stability measurement using the Ostell system
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 5 years
  Safety of MSC in patients. Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Gjerde, DDS, Principal Investigator — University of Bergen
Locations (1):
- Institute of Clinical Dentistry, University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gjerde C, Mustafa K, Hellem S, Rojewski M, Gjengedal H, Yassin MA, Feng X, Skaale S, Berge T, Rosen A, Shi XQ, Ahmed AB, Gjertsen BT, Schrezenmeier H, Layrolle P. Cell therapy induced regeneration of severely atrophied mandibular bone in a clinical trial. Stem Cell Res Ther. 2018 Aug 9;9(1):213. doi: 10.1186/s13287-018-0951-9. PMID 30092840